CLINICAL TRIAL: NCT06552793
Title: Evaluation of Post Extraction Hard Tissue Alteration Following Ridge Preservation In The Esthetic Zone Using Partially Demineralized Autogenous Dentine Graft Versus Xenograft: A Randomized Controlled Clinical Trial.
Brief Title: Post Extraction Alterations Following Ridge Preservation In The Esthetic Zone Using Partially Demineralized Autogenous Dentine Graft Versus Xenograft
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Riham Ahmad Alshiek Hani Alkurdee, principle investigator Riham Ahmad Master degree student, periodontology department, faculty of dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21524PER6-3-1
Record Dates: First submitted 2024-08-10; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Socket Preservation
Keywords: socket preservation; ridge preservation; autogenoues partially demineralized dentin graft; xenograft
MeSH Terms: interventions — Transplantation, Heterologous

STUDY DESIGN:
Intervention Model Description: A randiomized clinical trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autogenous partially demineralized dentin graft (Experimental): Following atraumatic tooth extraction, curettes will be used to remove granulation tissues, and the socket will be irrigated with sterile normal saline.Then the socket will be filled with Autogenous partially demineralized dentin graft (that will be prepared using tooth transformer device) followed by placement of a collagen membrane to cover the socket(The membrane will be shaped to extend 2-3 mm beyond the margins of the extraction socket and positioned just beneath the marginal mucosa) . Suturing technique will be a criss cross horizontal mattress to ensure that most of the grafting material is covered.
  Interventions: Biological: autogenous partially demineralized dentin graft
- Xenograft (Active Comparator): Following atraumatic tooth extraction, curettes will be used to remove granulation tissues, and the socket will be irrigated with sterile normal saline.Then the socket will be filled with xenograft graft followed by placement of a collagen membrane to cover the socket.( The membrane will be shaped to extend 2-3 mm beyond the margins of the extraction socket and positioned just beneath the marginal mucosa) Suturing technique will be a criss cross horizontal mattress to ensure that most of the grafting material is covered.
  Interventions: Biological: Xenograft

INTERVENTIONS:
Biological: autogenous partially demineralized dentin graft — tooth cleaning : form decay, tartar, soft tissue debris, fillings, cement then cut into fragments (5×5 mm) and inserted into the milling device (Tooth Transformer, Milan, Italy). A disposable box containing disposable liquid solutions will be inserted into the device to ensure the demineralization of the graft with 0.1 M hydrochloric acid, 10% hydrogen peroxide, and demineralized water as a wash.The decontamination of the granules will take place through UVA rays and ultrasounds, with temperature variations always lower than 43 ◦C to avoid damage to proteins. After 25 min, particle graft biomaterials will be obtained. The particles size will range from 815 µm with peaks up to 1110 µm.
  Arms: Autogenous partially demineralized dentin graft
Biological: Xenograft — Cortico-cancallous Bovine powder
  Arms: Xenograft

SUMMARY:
the aim of this study is to establish if there are clinical, radio-graphical and histomorphometrical differences between using Partially Demineralized Dentin graft versus Xenograft in the esthetic zone. as a clinical application in alveolar bone regeneration procedures related to implant dentistry, including socket preservation, alveolar ridge augmentation, after tooth extraction in the esthetic zone. After extraction of non-restorable teeth in the esthetic zone, will ridge preservation with application of partially demineralized autogenous dentin graft produce less hard tissue changes compared to xenograft?

The initial therapy consists of periodontal treatment (phase I therapy) including supragingival scaling, subgingival debridement if needed, adjustment of faulty restoration and polishing. The mechanical plaque control instructions for each patient include brushing and interdental cleaning techniques. Flapless and atraumatic tooth extraction will be initiated, Then the sockets will be carefully packed with the allocated graft material that are shaped to match the individual size and contours of each socket. Once the grafts are properly adapted to the sockets, they will be covered with collagen membrane. The membrane will be shaped to extend 2-3 mm beyond the margins of the extraction socket and positioned just beneath the marginal mucosa. To ensure its stability, a cross-suture will be performed, securing the membrane in place.

Intervention group: The socket will be filled with partially demineralized autogenous dentin graft Control group: The socket will be filled with xenograft . For both groups, All the subjects will be evaluated at pre-surgical, baseline and 6 months post surgical months for clinical parameters and baseline( immediate post-surgical and 6 months post-surgical . Outcomes: Change in radiographic horizontal ridge width at 1mm below the most coronal aspect of the crest , Change in radiographic horizontal ridge width at 3 and 5mm below the most coronal aspect of the crest,Change in radiographic buccal ridge height , Change in radiographic buccal ridge height ,Change in radiographic Palatal ridge height,Percentage of new vital bone formation,Percentage of residual bone graft,Implant Primary Stability.

Detailed Description: This study aims to evaluate clinical, radiographic and histomorphometrica

DETAILED DESCRIPTION:
The study aims to radiographically evaluate the dimentionsal changes of hard tissue after application of partailly deminerlized dentin graft verus xenograft in the esthatic zone .

Research Procedure in brief:

The study is to be conducted in the Oral Medicine and Periodontology department, Faculty of Dentistry- Cairo University, Egypt.Patients are to be selected from the outpatient clinic of the department of Oral Medicine and Periodontology, clinic of the department of Oral surgery and clinic of the department of Endodontics -Cairo University. The initial therapy consists of periodontal treatment (phase I therapy) including supragingival scaling, subgingival debridement if needed, adjustment of faulty restoration and polishing. The mechanical plaque control instructions for each patient include brushing and interdental cleaning techniques. surgical interventions: Atraumatic extraction.The patient will rinse their mouth with 0.12% Chlorhexidine Administration of 4% articaine hydrochloride with 1:100,000 epinephrine will be as local anesthetic agent.Flapless and atraumatic tooth extraction will be initiated, using 15C blade intrasulcular incision will be performed.A periotome will be utilized to sever the periodontal ligament (PDL) fibers, followed by extraction witha straight elevator and extraction forceps.

In the test group:

The autogenous partially demineralized dentin graft will be prepared as follows:

A high-speed fine finishing stone and saline irrigation will be used to clean the tooth and remove any decay, restoration, or foreign materials. Tooth will be rinsed twice in phosphate buffered saline. The tooth will be dried using air and ground with the Tooth Transformer device following the manufacturer's protocol. Dentin particles will be obtained with a dimension of 400 - 800 μm .

Preparation of the autogenous partially demineralized dentin matrix

* The extracted tooth will be cleaned with a diamond bur under abundant irrigation with physiological water. All filling materials (gutta-percha, composite, luting cements, etc.) will be removed with the outmost care and under magnification.
* Subsequently, the tooth will be cut into fragments (5 × 5 mm) and inserted into the milling device . According to the manufacturer, a disposable box containing disposable liquid solutions will be inserted into the device to ensure the demineralization of the graft with 0.1 M hydrochloric acid, 10% hydrogen peroxide, and demineralized water as a wash.
* The decontamination of the granules will take place through UVA rays and ultrasounds, with temperature variations always lower than 43 ◦C to avoid damage to proteins.
* After 25 min, particle graft biomaterials will be obtained. The particles size will range from 815 µm with peaks up to 1110 µm.
* All bone defects will be filled with the graft obtained from the TT grinder.
* Device for Tooth Processing (The Tooth Transformer TT):

Part 1: Tooth Cleaning After extraction, the tooth must be cleaned of tooth decay, tartar, soft tissue debris, fillings, cement, and prosthetic components. For the TT®, which calls for cutting the tooth into sections for the trituration stage .

Part 2: Tooth Grinding The TT® is equipped with a multipurpose sterilizable system that operates at low speed, which makes it possible to avoid the loss of tooth substance during pulverisation, despite the drawback of not being able to enter an entire tooth into the shredder .

Part 3: Treatment by Device The shredder is closed and inserted once the tooth has been placed. When the door is closed and the button is pressed, a liquid cartridge and a cylinder with a granulate collection cup (maker) are placed into the apparatus in their respective housings, the cartridge is activated by punching, and the procedure starts .

In control group:

Xenograft will be prepared in a separate room to keep patients blinded, where the allocated material will be administered 15 minutes after tooth extraction. A xenograft will be implanted in the alveolus.

Alveolar ridge preservation:

Following a thorough cleaning procedure,

Biopsy collection:

After 6 months healing a local anesthesia will be given, a full thickness mucoperiosteal flap will be detached in the augmented areas and a bone biopsy will be collected using a 4 mm trephine bur.

Implant placement:

After 6 months healing a local anesthesia will be given, a full thickness mucoperiosteal flap will be detached in the augmented areas an implant placement with sequences drill will be done.

Postoperative Care and follow up:

Participants will be given instructions to avoid any trauma to the operative site, refrain from interfering with the sutures, and to avoid consuming hot food or engaging in vigorous rinsing.

They will be encouraged to continue tooth brushing for the other parts of their dentition, while gentle tooth brushing for the operative site will be advised to be resumed after a two-week period.

Participants will be prescribed either Amoxicillin 500 mg (Misr Co. for Pharmaceutical Industries, Egypt) three times daily for seven days, or doxycycline 100 mg (Doxymycin, Nile Co. for Pharmaceuticals and Chemical Industries, Egypt) twice daily if they are sensitive to penicillin. In case of severe pain, Ibuprofen 600 mg (Brufen, Kahira Pharmaceuticals, Egypt) will be prescribed. To facilitate gentle rinsing, participants will be instructed to use a 0.12% Chlorhexidine mouthwash twice daily for a duration of two weeks .

The sutures will be removed two weeks after the surgery. On the first day postoperatively, a baseline cone-beam computed tomography (CBCT) scan will be conducted. A final follow-up visit and CBCT scan will be scheduled for six months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-restorable teeth and Type II extraction socket in the esthetic zone indicated for extraction for periodontal, carious or traumatic reasons.
* Healthy patients with adequate oral hygiene (bleeding on probing ≤20%; Plaque index ≤20%).
* Adult patients above 18 years old.
* Patients accept 6-months follow-up period and provide an informed consent.

Exclusion Criteria:

* Heavy smokers (more than 10 cigarettes per day or an electronic cigarette dose of >6 mg/ml of nicotine).
* Patients reporting systemic conditions that may compromise healing or bone metabolism (eg: diabetes).
* Patients with poor oral hygiene (bleeding on probing >20%; Plaque index >20%)
* The presence of acute periapical infection.
* The presence of severe periodontal destruction.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in radiographic horizontal ridge width | after 6 months postoperatively
  CBCT scans will be performed at baseline and 6 months postoperatively. Measurements will be taken at both time points using identical reference points and lines. To establish a reference, the most apical point of the extraction socket will be identified on the baseline image, and two reference lines will be drawn. The vertical reference line will be placed at the midpoint of the extraction socket, intersecting the apical reference point. Additionally, a horizontal reference line will be drawn perpendicular to the vertical line, passing through the apical reference point.The horizontal ridge width will be measured at three specific levels: 1 mm, 3 mm, and 5 mm below the most coronal aspect of the crest. These measurements will be denoted as HW-1, HW-3, and HW-5, respectively.

SECONDARY OUTCOMES:
Change in radiographic buccal and palatal ridge height: | after 6 months postoperatively.
  CBCT scans will be performed at baseline and 6 months postoperatively. Measurements will be taken at both time points using identical reference points and lines. To establish a reference, the most apical point of the extraction socket will be identified on the baseline image, and two reference lines will be drawn. The vertical reference line will be placed at the midpoint of the extraction socket, intersecting the apical reference point.
  The height of the alveolus will be measured at the midbuccal aspect (BH) and midlingual aspect (LH).
Percentage of new vital bone formation and residual graft | after 6 months postoperatively
  The biopsies will be stored in a 10% formalin solution for preservation.they will undergo decalcification in EDTA for a duration of four weeks. Following decalcification, the specimens will be processed and embedded in paraffin to create tissue blocks. Longitudinal sections of 5μm thickness will be cut from the paraffin blocks.stained using hematoxylin and eosin (H&E) or Masson's trichromatic (MT) stains for histological evaluation and histomorphometric analysis. Photomicrographs of the stained sections will be captured using a digital light microscope. Histomorphometric analysis will be performed to quantify the area percentage occupied by bone, graft particles, and soft tissue stroma relative to the total examined histological area using Image analyzer software.The software will be calibrated to automatically convert the measurement units produced by the program into actual micrometer units for accurate quantification.
Implant Primary Stability | after 6 months postoperatively
  The primary stability of the implant fixture will be assessed using the Osstell Mentor Resonance Frequency Analyzer (Osstell AB, Goteborg, Sweden). Two measurements will be taken in the buccolingual and mesiodistal directions for each implant. The average of these two measurements will be recorded as the representative implant stability quotient (ISQ) for each individual implant.

CONTACTS AND LOCATIONS:
Overall Officials: Manal M Hosny, Professor, Study Director — Cairo University; Weam A El-Battawy, Ass. Prof., Study Chair — Cairo University; Riham A Alshikh Hani Alkurdee, Bachelor, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt